CLINICAL TRIAL: NCT01167504
Title: Investigating the Formation of Salivary Films and How They Change in the Presence of Ingredients From Food and Oral Hygiene Products
Brief Title: Factors Controlling the Formation of Salivary Films
Acronym: SalFilm
Status: Completed | Type: Observational
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: IFR03-2010
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: saliva; food; sensory; oral health; film; pellicle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Saliva Sample Collection: Saliva collection
  Interventions: Other: Saliva sample collection

INTERVENTIONS:
Other: Saliva sample collection — Collection of either whole mouth saliva or parotid saliva. Whole mouth saliva is collected through stimulation by inert gum. Parotid saliva is collected by using a Lashley cup placed over the parotid duct and stimulated by a fruit sweet.
  Other Names: Whole mouth saliva; Parotid saliva

SUMMARY:
The aim of this study is to determine how different ingredients which are found in food and other consumer products affect the ability of saliva to form surface films.

Saliva forms a protective film on the surfaces inside the mouth. This film affects the way we consume and digest food and protects our teeth and other surfaces inside the mouth from disease and decay. It is not well known how this film forms, or which components in everyday life affect formation of the film, and therefore its protective properties.

Samples of saliva will be collected from apparently healthy volunteers. The properties of the film (thickness, density, strength, protein composition) will be studied in the laboratory under controlled conditions. The effects of common ingredients in foods and other products such as proteins, emulsifiers, preservatives and surfactants on the formation and properties of the film will be determined.

The results of this study will help us to understand how different ingredients can change the properties of saliva that may affect the way that we sense and digest food, and the ability of saliva to protect against decay and infection. This could, in the future lead to new ideas for developing:healthy foods (e.g. lower fat) that taste better, or more effective dental care products.

DETAILED DESCRIPTION:
The aim of this study is to determine the physical and biochemical mechanisms responsible for the formation and structure development (in vitro) of the salivary mucous film and the impact of common ingredients found in food or oral hygiene products.

Saliva forms a film or pellicle on oral surfaces which serves as a protective barrier and lubricates the oral tissues during food consumption. However, it also provides the primary site for bacterial attachment and the build up of plaque. Therefore the physical and molecular structure of the salivary film is important for how we sense and taste food, how food is broken down in the mouth, and its effectiveness as a protective barrier. Much is known about the composition of saliva, but very little is known about the composition and structure of the salivary film or pellicle. We believe that the film formation and its physical properties, such as viscosity and strength are the result of complex interactions between different proteins within saliva, and with other components such as calcium and other salts, food components such as proteins and emulsifiers, and active compounds found in oral hygiene products such as preservatives and surfactants. This study will determine how the salivary film forms, its molecular composition and which other critical components affect its ability to form a stable, protective barrier. This knowledge will hopefully, in the future contribute to strategies to design healthier foods and more effective oral hygiene treatments.

The physical properties of saliva are not stable as the proteins tend to aggregate following secretion, which affects the length of time the film formation can be studied (ex vivo). Therefore we need to use fresh human saliva samples collected from healthy volunteers using a defined protocol to ensure sample quality, and assess them within four hours of collection. Saliva will be collected (either whole mouth or parotid), taken to the laboratory and allowed to form films on model surfaces, representative of those found in the mouth. The rate of formation, strength, thickness and mass of the films will be studied using a range of physical methods. The protein content and composition will also be determined to identify the components responsible for various stages of film formation. Then, the influence of environmental conditions such as pH, calcium and salt will be determined. Finally, we will determine how the films interact with external components found in food and oral hygiene products such as proteins, emulsifiers, preservatives and surfactants. Although we are not studying the effects of dietary intervention on saliva properties, we want to determine the underlying mechanisms responsible for film formation and break down. Paired T-tests will be used to compare parotid with whole mouth saliva from the same volunteers. Two sample T-tests will be used for comparison of similar measurements on samples from different volunteers. Diagnostic checks on results will be performed to check whether transformations are required to meet normality assumptions.

Two types of saliva samples will be collected: Whole Mouth Saliva (WMS) and Parotid Saliva (PS). The saliva will be stored at 4ºC (WMS may also be centrifuged at 2700xg for 20 minutes at 5°C to remove aggregates) and used within 4 hours of collection, as protein aggregation begins immediately after secretion, affecting the film formation properties, as determined in previous work. A range of physical techniques will be employed to determine the rate and extent of film formation, as well as the thickness, mass and rheological properties, under the different solution conditions and in the presence and absence of added ingredients as described above. Protein concentration and composition will also be determined. This will enable improved experimental design (e.g. normalising protein concentration) to improve the quality of the results. The results will be used to inform the design of further studies with other centres of expertise in order to understand the impact on in vivo behaviour of the salivary film and, for example the sensory perception of foods and the role of saliva on digestion of food structures.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years old
* Gender:Male or Female
* nonsmokers

Exclusion Criteria:

* diabetics
* medical history of Tuberculosis or Hepatitis
* depressed or elevated blood pressure measurements (<90/50 or <95/50 if symptomatic or >160/100).
* take any medication which may affect saliva production
* are related to someone in the study team i.e. spouse, partner or immediate family member
* are pregnant, planning to become pregnant, or are currently breastfeeding.
* have results of the clinical screening which indicate, or are judged by the Human Nutrition Unit (HNU) Medical Advisor to be indicative of, a health problem which compromise the wellbeing of the volunteer if they participated, which would affect the study data.

In addition, prior to each sample donation, the following conditions will be checked, and volunteers will only be allowed to donate saliva if none of the following apply:

* They have any current dental or mouth problems (bleeding gums, sores on mouth, dry mouth syndrome)
* They have had a viral illness or chest infection within last 7 days
* They are not able to produce sufficient saliva
* Volunteers will be required to avoid eating and drinking (except water) for 1 hour prior to saliva collection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparently normal healthy volunteers from the local community able to donate saliva samples.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Wilde, PhD, Study Director — Quadram Institute Bioscience; Michael J Ridout, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between 16/6/2010 and 16/2/2012. A pool of 12 volunteers was required. 12 volunteers were recruited in 2010 and 2011, 3 further volunteers recruited in 2012 to replace 3 volunteers who left the study for personal reasons.
Pre-assignment Details: There were no significant events required following enrollment.
Groups:
- Saliva Sample Collection: Collection of whole mouth and parotid saliva samples
Period: Overall Study
Arm/Group | Saliva Sample Collection
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Volunteers were required to donate saliva for ex-vivo study, as described in protocol. A pool of 12 volunteers was maintained. 3 further volunteers had to be recruited following 3 losses due to personal reasons, i.e. not connected with study.
Groups:
- Saliva Sample Collection: Collection of whole mouth and parotid saliva
Arm/Group | Saliva Sample Collection
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15

OUTCOME MEASURES:

1. Primary Outcome: Impact of Ingredients on Thickness (Depth, nm) of Salivary Films Adsorbed Onto Solid Surfaces
Description: The principal output is to determine how ingredients in food and oral hygiene products affect the way that saliva forms films on surfaces similar to those found inside the mouth. We will determine the main physical properties of the film such as thickness (nm), adsorbed mass (ng/cm^2), density (ng/cm^3) measured by adsorbing whole mouth saliva onto solid silica surfaces and measuring the above properties of the film using Dual Polarisation Interferometry and a Quartz Crystal Microbalance. The effect of ingredients from food and oral hygiene products on the above measured parameters will be determined.
Time Frame: Within 4 hours of saliva collection.
Population: Based on published results of saliva pellicle thickness, power calculations showed that 12 individuals would provide sufficient statistical significance to determine the effect of added ingredients on salivary film thickness.
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Saliva Sample Collection
Number analyzed (Participants) | 12
nm | 27 (8)

2. Secondary Outcome: Defined Behaviour of Salivary Film Formation
Description: A secondary output is a well defined description of the film formation behaviour of "normal"saliva in terms of thickness (nm), viscoelastic modulus (mN/m) and temporal behaviour. This will be used to develop model or artificial salivas saliva that forms films in the same way as real saliva ex vivo, that can be used to screen the effects of different compounds and ingredients, without having to collect fresh saliva from human volunteers. The measure is the rate of increase in film thickness (depth, nm) as a function of time, measured by adsorbing whole mouth saliva onto a solid silica surface and measuring the film thickness using Dual Polarisation Interferometry and Quartz Crystal Microbalance.
Time Frame: Within 4 hours of saliva collection.
Population: Literature data and power calculations were used to calculate the number of individuals required to show a statistical significant effect of the presence of ingredients on the thickness of the salivary film.
Measure: Mean (Standard Deviation); unit: nm/cm2/min
Arm/Group | Saliva Sample Collection
Number analyzed (Participants) | 12
nm/cm2/min | 868 (475)

ADVERSE EVENTS:
Arm/Group | Saliva Sample Collection
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
No adverse events were reported. The number of volunteers required gave acceptable statistics as anticipated. The study was completed on time

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes